CLINICAL TRIAL: NCT02690402
Title: Fragility Multidisciplinary Evaluation and Adapted Physical Activity
Brief Title: Fragility and Adapted Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-PP-12
Record Dates: First submitted 2015-10-05; First posted 2016-02-24 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Fragility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adapted physical activity (Experimental): a personalized care will be offered in terms of adapted physical activity
  Interventions: Behavioral: adapted physical activity

INTERVENTIONS:
Behavioral: adapted physical activity — The study begins with an evaluation of physical strenght and cognitive and psychometric assessment.Then, a personalized care will be offered in terms of adapted physical activity. The evaluation protocol will be performed again to measure the impact of physical activity three months after the first assessment.

SUMMARY:
Older people are a very heterogeneous population characterized by a high interindividual variability. Functional abilities (walking, transfers ...) used to classify individuals aged (Lalive d'épinay et al., 1999) in three categories: independent, frail and dependent (HAS, 2005). Frailty is generally considered as a state that precedes dependent status and, unlike the latter, is still reversible (Fried et al., 2001). Now, it's necessary to understand and quantify the indicators above the dependence of the elderly from a multidisciplinary approach to frailty, is a critical public health issue for developing non-drug therapeutic interventions adapted to delay the institutionalization. Through this study, it is to identify risk and protective factors of frailty and their relationships with physical activity, evaluate them and propose an appropriate care to the patient. This study should enable the production of new scientific knowledge to improve the health and quality of life of older people.

DETAILED DESCRIPTION:
Older people are a very heterogeneous population characterized by a high interindividual variability. Functional abilities (walking, transfers ...) used to classify individuals aged (Lalive d'épinay et al., 1999) in three categories: independent, frail and dependent (HAS, 2005). Frailty is generally considered as a state that precedes dependent status and, unlike the latter, is still reversible (Fried et al., 2001). These authors proposed criteria: physical inactivity (low levels of physical activity), unintentional weight loss (more than 5% of body weight over 6 months), perceived general fatigue, weakness of grip strength (handgrip) and slow speed walk. Nevertheless, at present, other more objective evaluation methods that include mobility, balance, muscle strength, endurance and cognition are necessary. Furthermore, psychological characteristics have not been studied with frailty indicators, except to walk speed. Now, these last are important levers of people adherence to physical activity programs (Baert et al., 2011). In this sense, better understand and quantify the indicators above the dependence of the elderly from a multidisciplinary approach to frailty, is a critical public health issue for developing non-drug therapeutic interventions adapted to delay the institutionalization.

The proposed study is to items (a) to characterize the functional dimensions of frailty from objective indicators and (b) putting them in relation to the cognitive and psychosocial characteristics of the elderly in order to define individual devices of care through physical activity.

To meet these objectives, it is necessary to include a large number of people in a comprehensive evaluation protocol physical, and their psycho-social and cognitive characteristics.

The research will begin with an inclusive visit by a medical doctor. Evaluation begins with a impedancemetric measurement, followed by posturographic evaluation. Then, in a first phase, patients will perform walk tests (e.g., 6 minutes, 10 m) during which spatiotemporal parameters of gait cycle, and the electromyographic activity of the different muscles of the lower limbs will be quantified. After the walk test, each subject will receive an evaluation of the strength of the ankle and knee muscles by an isokinetic dynamometer. During these contractions, the surface electromyographic activity of patients will also be recorded. In a second phase, subjects will perform a series of repetitions at 50% of maximum voluntary contraction (MVC) on the isokinetic dynamometer, to measure strength endurance. Thirdly, participants will be asked to complete cognitive tests and psychometric questionnaires. Finally, a personalized care will be offered in terms of adapted physical activity. The evaluation protocol will be performed again to measure the impact of physical activity three months after the first assessment.

Through this assessment, it is to identify risk and protective factors of frailty and their relationships with physical activity, evaluate them and propose an appropriate care to the patient. This study should enable the production of new scientific knowledge to improve the health and quality of life of older people.

ELIGIBILITY:
Inclusion Criteria:

* Patient who signed the informed consent
* Older men and women ≥ 65 years
* Can walk without technical help

Exclusion Criteria:

* Patient with protective measures (guardianship, curatorship, and deprivation of liberty).
* Patient with a neurological problem
* No affiliation to a social security scheme (beneficiary or assignee)
* Knee and / or hip prosthesis
* Orthopedic complications with repercussions on walking activities

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 970 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Gait analysis | change from baseline physical activity at 3 months
Isocinetic evaluation | change from baseline physical activity at 3 months
Questionnaire : Physical activity, psychometric | change from baseline physical activity at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GUERIN, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided